CLINICAL TRIAL: NCT04495790
Title: Advanced Integrative Oncology Treatment for Adult and Pediatric Patients With Cancer: A Prospective Outcomes Study
Brief Title: AIMS Cancer Outcomes Study
Acronym: ACOS
Status: Recruiting | Type: Observational
Sponsor: Advanced Integrative Medical Science Institute (Other)
Responsible Party: Sponsor
Other Study IDs: ACOS
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2023-01

CONDITIONS: Neoplasms; Neoplasm Malignant; Advanced Cancer; Advanced Solid Tumor; Oncology
Keywords: Integrative Oncology; Naturopathic Oncology; Phytomedicine; Metabolic Therapy; Immunotherapy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The overall aim is to describe disease-free survival (DFS) in early stage cancer patients and three-year overall survival (OS) outcomes in advanced stage cancer patients receiving Advanced Integrative Oncology (AIO) treatment in a prospective consecutive case series outcomes study. We will collect data and study outcomes for patients with cancer who receive care at AIMS Institute.

DETAILED DESCRIPTION:
It is estimated that between 50 and 80% of cancer patients in the United States (US) supplement their conventional medical treatment regimen with some form of complementary or alternative medicine (CAM) therapy or practice. A smaller percentage of these patients receive medical treatment from naturopathic doctors (NDs) who are board certified in naturopathic oncology (Fellows of the American Board of Naturopathic Oncology, FABNO) or have equivalent experience in caring for cancer patients. This level of care is being defined here as Advanced Integrative Oncology (AIO). AIO clinics provide comprehensive science- and experience-based naturopathic medical oncology integrated with the individual patient's conventional medical treatment.

Although there have been some studies of alternative and complementary medicine use by both adult and pediatric cancer patients, little is known about the effectiveness of naturopathic medicine provided to patients with cancer in an integrative setting. Increasing numbers of parents of children seek out naturopathic physicians and other integrative oncologists for evidence-based complementary integrative therapy that is coordinated with the child's standard oncology treatment plan. The AIMS Institute provides nutritional and botanical medicine care to children with leukemia, brain cancer, and osteosarcoma. Despite the widespread use of integrative oncology by children with cancer, little is known about the effectiveness of these therapies in pediatric cancer patients.

While there is scientific evidence supporting specific treatments that are commonly used, systematic study of their effectiveness, especially when used in combination as commonly recommended, is sparse. We believe that an early step in the evaluation of clinical outcomes associated with CAM is to take a health services approach and seek to answer the question: "Does exposure to AIO services improve the clinical outcomes of patients with cancer?"

ELIGIBILITY:
Inclusion Criteria:

1. A new patient coming in for a first office call (FOC) or first consultation via telemedicine with a diagnosis of cancer, or
2. An established patient with a diagnosis of cancer receiving treatment at the AIMS Institute;
3. If over 18 years of age are able to understand study design adequately and provide signed informed consent (IC) to enrollment;
4. If younger than 18 years of age informed assent from the child and informed consent from a parent or guardian who is able to understand the study design adequately and provide signed informed consent for the pediatric patient;
5. A confirmed diagnosis of cancer based on medical oncology medical records.

Exclusion Criteria:

1. Patients not diagnosed with cancer;
2. Telehealth patients;
3. Cannot read or understand English well enough to read and sign the consent form and complete the questionnaires;
4. Unwilling to participate in the AIMS Institute observational study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All cancer patients who seek care at AIMS Institute and meet inclusion/exclusion criteria are eligible to participate in this study. Participants will be informed and educated about the prospective outcomes study by clinical staff as part of patient registration and the clinical intake process. Patients may be referred to AIMS Institute by cancer care centers, oncologists and other health care providers, or patients may be self-referred.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-18 (Actual); Primary Completion 2025-05-18 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
AIM 1 (survival) | 5 Years
  Measure DFS and OS in advanced stage cancer patients who receive AIO treatments at AIMS Institute.

SECONDARY OUTCOMES:
AIM 2 (treatment) | 5 Years
  Describe AIO treatments prescribed and provided by AIMS physician and their medical staff.
AIM 3 (correlate survival with treatment) | 5 Years
  Correlate survival outcomes with treatments received.

CONTACTS AND LOCATIONS:
Locations (1):
- AIMS Institute, Seattle, Washington, United States

REFERENCES:
- [Background] Ladas EJ. Integrative Medicine in Childhood Cancer. J Altern Complement Med. 2018 Sep/Oct;24(9-10):910-915. doi: 10.1089/acm.2018.0224. PMID 30247963
- [Background] Neuhouser ML, Patterson RE, Schwartz SM, Hedderson MM, Bowen DJ, Standish LJ. Use of alternative medicine by children with cancer in Washington state. Prev Med. 2001 Nov;33(5):347-54. doi: 10.1006/pmed.2001.0911. PMID 11676573
- [Background] Ghiasuddin A, Wong J, Siu AM. Complementary and alternative medicine practices, traditional healing practices, and cultural competency in pediatric oncology in Hawai' i. J Integr Med. 2016 Sep;14(5):374-9. doi: 10.1016/S2095-4964(16)60267-6. PMID 27641608
- [Background] Lerman C, Trock B, Rimer BK, Jepson C, Brody D, Boyce A. Psychological side effects of breast cancer screening. Health Psychol. 1991;10(4):259-67. doi: 10.1037//0278-6133.10.4.259. PMID 1915212
- [Background] McHorney CA, Ware JE Jr, Lu JF, Sherbourne CD. The MOS 36-item Short-Form Health Survey (SF-36): III. Tests of data quality, scaling assumptions, and reliability across diverse patient groups. Med Care. 1994 Jan;32(1):40-66. doi: 10.1097/00005650-199401000-00004. PMID 8277801
- [Background] Seely D, Wu P, Fritz H, Kennedy DA, Tsui T, Seely AJ, Mills E. Melatonin as adjuvant cancer care with and without chemotherapy: a systematic review and meta-analysis of randomized trials. Integr Cancer Ther. 2012 Dec;11(4):293-303. doi: 10.1177/1534735411425484. Epub 2011 Oct 21. PMID 22019490
- [Background] Ma Y, Chapman J, Levine M, Polireddy K, Drisko J, Chen Q. High-dose parenteral ascorbate enhanced chemosensitivity of ovarian cancer and reduced toxicity of chemotherapy. Sci Transl Med. 2014 Feb 5;6(222):222ra18. doi: 10.1126/scitranslmed.3007154. PMID 24500406
- [Background] McCulloch M, Broffman M, van der Laan M, Hubbard A, Kushi L, Abrams DI, Gao J, Colford JM Jr. Colon cancer survival with herbal medicine and vitamins combined with standard therapy in a whole-systems approach: ten-year follow-up data analyzed with marginal structural models and propensity score methods. Integr Cancer Ther. 2011 Sep;10(3):240-59. doi: 10.1177/1534735411406539. Epub 2011 Sep 30. PMID 21964510
- [Background] Pierce JP, Stefanick ML, Flatt SW, Natarajan L, Sternfeld B, Madlensky L, Al-Delaimy WK, Thomson CA, Kealey S, Hajek R, Parker BA, Newman VA, Caan B, Rock CL. Greater survival after breast cancer in physically active women with high vegetable-fruit intake regardless of obesity. J Clin Oncol. 2007 Jun 10;25(17):2345-51. doi: 10.1200/JCO.2006.08.6819. PMID 17557947